CLINICAL TRIAL: NCT05906511
Title: Pharmacokinetics and Pharmacodynamics of Oral and Vaporized Delta-9-Tetrahydrocannabinol (THC) in Older Adults
Brief Title: PK/PD of Oral and Vaporized Delta-9-Tetrahydrocannabinol (THC) in Older Adults
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Joao De Aquino, Assistant Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2000035354; 1R21DA057240-01 (NIH)
Record Dates: First submitted 2023-05-25; First posted 2023-06-18 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Pain, Tolerance; Oral vs Vaporized THC; Abuse Liability
Keywords: Pharmacokinetics THC; Pharmacodynamics THC
MeSH Terms: conditions — Pain | interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: This is a double-blind, placebo-controlled, crossover study, randomizing 20 men and women aged 65 years or older to two doses of oral THC and vaporized THC.
Who Masked: Participant, Investigator
Masking Description: Study medication will be prepared by study pharmacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Dronabinol 5mg (Active Comparator): Dronabinol 5 mg
  Interventions: Drug: Dronabinol 5 MG
- Dronabinol 10mg (Placebo Comparator): Dronabinol 10 mg
  Interventions: Drug: Dronabinol 10 MG
- Vaporized THC 2mg (Active Comparator): Vaporized THC 2mg
  Interventions: Drug: 2mg Purified THC in an ethanolic solution
- Vaporized THC 4mg (Active Comparator): Vaporized THC 4 mg
  Interventions: Drug: 4mg Purified THC in an ethanolic solution
- Placebo (Placebo Comparator): Masked oral placebo or vaporized saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol 5 MG — Dronabinol 5 mg
  Other Names: "Marinol"
  Arms: Dronabinol 5mg
Drug: Dronabinol 10 MG — Dronabinol 10mg
  Other Names: "Marinol"
  Arms: Dronabinol 10mg
Drug: 2mg Purified THC in an ethanolic solution — 2mg Purified THC in an ethanolic solution
  Arms: Vaporized THC 2mg
Drug: 4mg Purified THC in an ethanolic solution — 4mg Purified THC in an ethanolic solution
  Arms: Vaporized THC 4mg
Drug: Placebo — Oral placebo and/or vaporized saline
  Arms: Placebo

SUMMARY:
The overarching goal of this double-blind, placebo-controlled, crossover study is to characterize the pharmacokinetic (PK) and pharmacodynamic (PD) effects of the main analgesic and psychoactive constituent of cannabis, delta-9 tetrahydrocannabinol (THC), among older adults - the fastest growing population of cannabis consumers, and the most likely age cohort to use cannabinoids to relieve pain. This protocol includes two sub-studies, each randomizing 20 men and women aged 65 years or older to receive two administration routes of THC; oral administration and vaporized administration.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, crossover study, with two sub-studies each focusing on different routes of THC administration.

Oral THC Sub-Study: 20 men and women aged 65 years or older, will be randomized to two doses of oral THC (5 mg and 10 mg). Across three, 8-hour test sessions, participants will receive a random sequence of 3 conditions: 5 mg oral THC; 10 mg oral THC; oral placebo.

Vaporized THC Sub-Study: 20 men and women aged 65 years or older will be randomized to two doses of vaporized THC (2 mg and 4 mg). Across three 8-hour test sessions, participants will receive a random sequence of 3 conditions: 2 mg vaporized THC; 4 mg vaporized THC; and vaporized placebo.

For both the Oral and Vaporized THC Sub-Studies, blood samples will be regularly collected from an intravenous line, up to 8 hours post-dose, and at 24 hours post-dose, to assess the PK of THC and its phase I and II metabolites. PD effects of THC on pain will be measured with Quantitative Sensory Testing (QST), a psychophysical technique used to reliably measure pain sensitivity and investigate pain modulatory mechanisms. The abuse liability of THC will be measured using an established drug reinforcement paradigm. General adverse, cardiovascular, and cognitive/psychomotor effects of THC will be thoroughly assessed with behavioral, physiological, and neuropsychological methods.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female participants aged 65 ≥ years old
2. Prior exposure to THC or cannabis least once in the last 10 years; 1-10 times in the last 20 years; or more than 20 times in their lifetime
3. Capable of providing informed consent in English.

Exclusion Criteria:

1. Meeting DSM-5 criteria for psychiatric/substance use disorders (SUD) other than tobacco use disorder, within the last year
2. Current use of cannabinoid products, as evidenced by a urine drug screen
3. Having a history of treatment for cannabis use disorder
4. History of intent or current intent of abstaining from cannabis use
5. Clinically significant medical disorders (e.g. liver/kidney dysfunction, immunosuppressing conditions, history or presence of epilepsy, seizures, head trauma with loss of consciousness)
6. Medical conditions that increase the risk of respiratory problems (e.g. COPD, asthma, recuring bronchitis, reactive airway disorder)* (does not apply to the Oral THC Sub-Study)
7. History of environmental sensitivities (e.g. bronchospastic allergies, multiple chemical sensitivities) or other airway sensitivities that require the use of an epi pen*(does not apply to the Oral THC Sub-Study)
8. Neurological conditions that may change the response to nociceptive stimuli (e.g., stroke, neuropathy), or that lead to loss of balance, evidenced by a neuro-sensory exam
9. Contraindications for exposure to nociceptive stimuli, such as untreated hypertension
10. Current regular use of drugs known to affect pain, or that are prominent inducers or inhibitors of CYP2C9, CYP3A4, or UGTA19 (e.g., carbamazepine, valproate, fluvoxamine, and paroxetine)
11. Major neurocognitive disorders precluding participation, evidenced by a clinical exam
12. Abnormal EKG, arrythmia, vasospastic disease, chronic heart failure, or presence of a pacemaker
13. Elevation of liver enzymes (ALT, AST) 2x the normal limit or higher
14. Personal or family history of primary psychotic disorders, or mood disorders with psychotic features
15. Current suicidal ideation
16. Allergy or serious adverse reactions to sesame oil, THC, or cannabis
17. Having received any drug as part of a research study within 30 days prior to receiving the study medication in the current study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Peak concentration (Cmax) | Up to 8 hours
  Serial blood samples will be collected for plasma levels of THC; its phase I metabolite 11-hydroxy-THC (OH-THC); phase II metabolite 11-nor-9-carboxy-THC (THC-COOH); and THC-COOH glucuronide. For THC and all other analytes, the peak concentration (Cmax) will be derived using a linear noncompartmental analysis.
Time to attain Cmax concentration (Tmax) | Up to 8 hours
  Serial blood samples will be collected for plasma levels of THC; its phase I metabolite 11-hydroxy-THC (OH-THC); phase II metabolite 11-nor-9-carboxy-THC (THC-COOH); and THC-COOH glucuronide. For THC and all other analytes, the time to attain Cmax concentration (Tmax) will be derived using a linear noncompartmental analysis.
Area under the plasma concentration-time curve (AUC0-8h) | Up to 8 hours
  Serial blood samples will be collected for plasma levels of THC; its phase I metabolite 11-hydroxy-THC (OH-THC); phase II metabolite 11-nor-9-carboxy-THC (THC-COOH); and THC-COOH glucuronide. For THC and all other analytes, the area under the plasma concentration-time curve (AUC0-8h) will be derived using a linear noncompartmental analysis.
Nociception | Up to 8 hours
  Multimodal quantitative sensory testing (QST) will be used ensure that various types of afferent fibers are engaged, so that the analgesic efficacy of THC can be comprehensively investigated. A composite pain sensitivity measure as a Z-score (ranging from -1 to +1) will be derived from the QST battery, with greater scores indicating a higher sensitivity to pain.
Abuse Liability | Up to 8 hours
  A modified Multiple-Choice Procedure (MPC) will be used to measure abuse liability. The MCP was developed and validated by Roland Griffiths to efficiently assess drug reinforcement - including cannabinoid-induced reinforcement. In each of the 6 experimental sessions, participants will choose between forfeiting or receiving escalating sums of money, on a scale of values between -$20.00 and $20.00; or re-receiving the study medication assigned for that day. The primary outcome will be the crossover point, the value at which the participant chooses money rather than the study medication, which will be determined for each session.

CONTACTS AND LOCATIONS:
Overall Officials: Joao P. De Aquino, M.D., Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaskie B, Ayyagari P, Milavetz G, Shane D, Arora K. The Increasing Use of Cannabis Among Older Americans: A Public Health Crisis or Viable Policy Alternative? Gerontologist. 2017 Nov 10;57(6):1166-1172. doi: 10.1093/geront/gnw166. PMID 28077451
- [Background] Solomon HV, Greenstein AP, DeLisi LE. Cannabis Use in Older Adults: A Perspective. Harv Rev Psychiatry. 2021 May-Jun 01;29(3):225-233. doi: 10.1097/HRP.0000000000000289. PMID 33660625
- [Background] Mahvan TD, Hilaire ML, Mann A, Brown A, Linn B, Gardner T, Lai B. Marijuana Use in the Elderly: Implications and Considerations. Consult Pharm. 2017 Jun 1;32(6):341-351. doi: 10.4140/TCP.n.2017.341. PMID 28595684
- [Background] Gagliese L. What do experimental pain models tell us about aging and clinical pain? Pain Med. 2007 Sep;8(6):475-7. doi: 10.1111/j.1526-4637.2007.00360.x. No abstract available. PMID 17716320
- [Background] Moore AR, Clinch D. Underlying mechanisms of impaired visceral pain perception in older people. J Am Geriatr Soc. 2004 Jan;52(1):132-6. doi: 10.1111/j.1532-5415.2004.52023.x. PMID 14687328
- [Background] Lautenbacher S, Kunz M, Strate P, Nielsen J, Arendt-Nielsen L. Age effects on pain thresholds, temporal summation and spatial summation of heat and pressure pain. Pain. 2005 Jun;115(3):410-418. doi: 10.1016/j.pain.2005.03.025. PMID 15876494
- [Background] Backonja MM, Attal N, Baron R, Bouhassira D, Drangholt M, Dyck PJ, Edwards RR, Freeman R, Gracely R, Haanpaa MH, Hansson P, Hatem SM, Krumova EK, Jensen TS, Maier C, Mick G, Rice AS, Rolke R, Treede RD, Serra J, Toelle T, Tugnoli V, Walk D, Walalce MS, Ware M, Yarnitsky D, Ziegler D. Value of quantitative sensory testing in neurological and pain disorders: NeuPSIG consensus. Pain. 2013 Sep;154(9):1807-1819. doi: 10.1016/j.pain.2013.05.047. Epub 2013 Jun 3. PMID 23742795
- [Background] Griffiths RR, Troisi JR, Silverman K, Mumford GK. Multiple-choice procedure: an efficient approach for investigating drug reinforcement in humans. Behav Pharmacol. 1993 Feb;4(1):3-13. PMID 11224166